CLINICAL TRIAL: NCT02795663
Title: Deep Brain Stimulation and Parkinson's Disease: Analysis of the Modifications of the Cortical Activation During Driving Tasks and During Tasks Involving the Control of the Impulses by Means of the Optical Imaging and of the Technique of Delay Discounting Task
Brief Title: Deep Brain Stimulation and Parkinson's Disease
Acronym: SCP TCI NIRS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2013_843_0016
Record Dates: First submitted 2016-05-26; First posted 2016-06-10 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
Keywords: Near-InfraRed Spectroscopy (NIRS); Deep brain stimulation of SubThalamic Nucleus (DBS)
MeSH Terms: conditions — Parkinson Disease

ARMS (3):
- parkinson's patient stimulated at STN level (Experimental): 15 parkinson's disease patients stimulated at STN level NIRS EEG HR recording
  Interventions: Device: NIRS EEG HR recording
- non STN (Experimental): 5 Parkinson's Disease patients who received stimulation in another target that the STN NIRS EEG HR recording
  Interventions: Device: NIRS EEG HR recording
- control (Experimental): 20 control patients undergoing DBS for the treatment of OCD NIRS EEG HR recording
  Interventions: Device: NIRS EEG HR recording

INTERVENTIONS:
Device: NIRS EEG HR recording — NIRS EEG HR recording

SUMMARY:
* Background : Deep brain stimulation of SubThalamic Nucleus (STN-DBS) is an effective treatment for a large variety of movement disorders. However, the efficacy of STN-DBS relies on unclear mechanisms.
* Purpose: In this study, using optical imaging, the investigators will evaluate the cortical hemodynamic changes induced by STN-DBS of parkinsonian patients during motor task and delay discounting task. the investigators will perform an optical imaging study using Near-InfraRed Spectroscopy (NIRS) in a parkinsonian patient after STN-DBS. The investigators will measure bilateral local cortical hemodynamic changes under "On" and "Off" stimulation conditions and during a motor task (left hand movement) and delay discounting task Relative concentration changes of oxy-Hb, deoxy-Hb, and total Hb will be continuously analyze.
* Primary outcome: Study of local cortical hemodynamic change (oxy-Hb, deoxy-Hb, and total Hb) under " on " and " off " stimulation during a motor task.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting Parkinson disease and treated by STN-DBS.
* For comparison patients: Patients treated by DBS in other target.

Exclusion Criteria:

* Patients who cannot be treated by DBS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Study of local cortical hemodynamic change (oxy-Hb, deoxy-Hb, and total Hb) | 1 month,
  under " on " and " off " stimulation during a motor task.

SECONDARY OUTCOMES:
Study of local cortical hemodynamic change (oxy-Hb, deoxy-Hb, and total Hb) | 1 month
  under " on " and " off " stimulation during delay discounting task.
Study of QUIP score (QUIP scale) | 3 month
Comparison of local cortical hemodynamic changes (oxy-Hb, deoxy-Hb, and total Hb) with the localisation of the contact use for STN-DBS stimulation | 1 month
  between patient with ICD and patient without ICD
Comparison of local cortical hemodynamic changes (oxy-Hb, deoxy-Hb, and total Hb) with intensity of STN-DBS stimulation | 1 month
Study of local cortical hemodynamic changes (oxy-Hb, deoxy-Hb, and total Hb) with intensity of NonSTN-DBS stimulation | 1 month
  under " on " and " off " stimulation during a motor task and a delay discounting task (in order to obtain a qualitative comparison between GPi-DBS and STN-DBS.
Study of delayed discounting task (DDT) score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel LEFRANC, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Result] Mahmoudzadeh M, Wallois F, Tir M, Krystkowiak P, Lefranc M. Cortical hemodynamic mapping of subthalamic nucleus deep brain stimulation in Parkinsonian patients, using high-density functional near-infrared spectroscopy. PLoS One. 2021 Jan 25;16(1):e0245188. doi: 10.1371/journal.pone.0245188. eCollection 2021. PMID 33493171